CLINICAL TRIAL: NCT03393832
Title: Oral Care: An Important Adjunctive Therapy to Improve Feeding Tolerance in Infants With Gastroschisis
Brief Title: Oral Care in Infants With Gastroschisis
Status: Active, not recruiting | Type: Observational
Sponsor: Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, Amy Hair, Assistant Professor, Baylor College of Medicine
Other Study IDs: H41227
Record Dates: First submitted 2018-01-03; First posted 2018-01-09 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-02

CONDITIONS: Gastroschisis
Keywords: Oral care; Oropharyngeal mother's milk
MeSH Terms: conditions — Gastroschisis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Stools will be collected daily for 1st week of life then weekly for 3 weeks to study the intestinal microbiome and relative abundance of various bacteria. Oral care samples (mother's own milk) will be collected at time of stool collection to characterize/compare the abundance of bacteria in the oral care vs stool samples. Saliva will be collected to identify/quantify salivary gland proteins at these times: baseline sample following study enrollment (0-72 hours), before surgical closure of gastroschisis, daily from DOL 10 to when infant reaches full enteral feeds (140 cc/kg/day), and one after infant reaches full enteral feeds. Collected samples will be stored in the Neonatal Nutrition Research Biorepository.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Oral Care with Mother's Milk: All infants admitted to the Texas Children's Hospital NICUs who have mother's milk available will receive oral care with mother's milk.
- Oral Care with Sterile Water: Infants will receive oral care with sterile water when mother's milk is not available.

SUMMARY:
Gastroschisis is a rare abdominal wall defect. Though survival rate is high, there are significant complications related to feeding intolerance and infections. Recently, oral care with breast milk has been studied in extremely premature infants and has been shown to improve both feeding tolerance and protect against infection. Though only studied in premature infants, it is likely that other populations of patients can benefit form oral care as well. This is a prospective observational cohort study looking at infants with gastroschisis admitted to the Texas Children's Hospital Newborn Center NICU (level II and level IV) who receive oral care with mother's milk or sterile water when mother's milk is not available. The study is aimed to demonstrate the benefits of oral care with breast milk in infants with gastroschisis. Additionally, the investigators will evaluate how oral care with breast milk affects the intestinal bacterial environment and how oral care with breast milk affects the secretion of certain proteins from the salivary gland.

Primary hypothesis: The primary objective is to compare the magnitude of increase in intestinal microbiota alpha diversity over a four week period between infants who receive oral care with mother's milk and those receiving oral care with sterile water using a paired analysis.

Secondary hypothesis:

* Oral care with breast milk will decrease the days to start enteral feeds after primary surgical closure inpatients with gastroschisis.
* Oral care with breast milk will decrease the days to reach full enteral feeds of 140 cc/kg/day in patients with gastroschisis.
* Oral care with breast milk will decrease length of stay in patients with gastroschisis.
* Oral care with breast milk will increase secretion of certain proteins, such as vascular endothelial growth factor, from the salivary gland.

DETAILED DESCRIPTION:
Breast milk is recommended for most infants by the American Academy of Pediatrics as there are multiple benefits. However, some infants, such as extremely premature infants, are unable to receive enteral nutrition for a variety of clinical reasons. In order provide these infants with some of the benefits of mother's milk, a novel adjunctive therapy called oral care has been developed. Oral care consists of applying mother's breast milk to the buccal mucosa. Oral care has been studied in the premature infant population and been shown to improve both feeding tolerance and to provide immune protection. Although only studied in the premature population, many institutions including Texas Children's Hospital have adopted oral care as a standard of care for all infants as oral care poses minimal risk to the patient and has many potential benefits. Gastroschisis is a rare abdominal wall defect. Although the survival rate for infants with gastroschisis is high, there are significant morbidities related to feeding intolerance and infection. The investigators believe that this population of patients will also benefit from oral care.

The mechanism by which oral care works is not completely understood. It is theorized that oral care stimulates the oropharyngeal-lymphoid tissue in the buccal mucosa. Additional mechanisms include alteration of the intestinal microbiome. The intestinal microbiome is the millions of microorganisms that line the intestine. Normally, there is a mutually beneficial relationship. The intestinal microbiome is altered by many factors, including gestational age, antibiotic use, type of delivery, etc. Alterations in the microbiome can be detrimental and cause severe diseases such as necrotizing enterocolitis. Thus, far studies have shown that oral care alters the oral microbiome to include more healthy bacteria. The investigators believe that oral care with breast milk will be associated with a more diverse fecal microbiota. Finally, the investigators will evaluate a novel mechanism by which the investigators believe oral care is protective; via increased salivary gland secretion of certain proteins important for healing. In particular, saliva contains vascular endothelial growth factor, which is important for palatal wound healing and alimentary tract healing.

ELIGIBILITY:
Inclusion Criteria:

• Infants with a primary diagnosis of gastroschisis

Exclusion Criteria:

* Gestational age less than 30 weeks
* Birth weight less than 1,000 g
* Other major congenital anomalies or clinically significant heart disease
* First dose of oral care greater than 72 hours after birth
* Early transfer to another institution

Max Age: 3 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Infants with a diagnosis of gastroschisis are identified either prenatally through the Texas Children's Hospital Fetal Center or upon admission to the Texas Children's Hospital Neonatal Intensive Care Unit (NICU).
Sampling Method: Non-Probability Sample
Enrollment: 27 (Actual)
Dates: Start 2017-10-14 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Microbiome Outcome | 4 weeks
  The primary objective is to compare the magnitude of increase in intestinal microbiota alpha diversity over a four week period between infants who receive oral care with mother's milk and those receiving oral care with sterile water using a paired analysis.

SECONDARY OUTCOMES:
Days to start enteral feeds after primary surgical closure between the two cohorts | The current average time to start feeds after surgical closure is 15 days.
  The first secondary objective is to compare the days to start enteral feeds after primary surgical closure between the two cohorts.
Days to reach full enteral feeds of 140 cc/kg/day between the two study cohorts | The current average time to reach full enteral feeds is 105 days.
  The second secondary objective is to compare days to reach full enteral feeds of 140 cc/kg/day between the two study cohorts.
Length of stay between the two study cohorts | The current average length of stay is 70 days.
  The third secondary objective is to compare length of stay between the two study cohorts.
Salivary Gland Outcome: levels of salivary proteins between the two study cohorts | The average is 6 weeks.
  The final secondary objective is to compare levels of salivary proteins between the two study cohorts from birth to when infant achieves full enteral feeds of 140 cc/kg/day, using either ELISA or Luminex Mulitplex assays.

CONTACTS AND LOCATIONS:
Overall Officials: Amy B Hair, MD, Principal Investigator — Baylor College of Medicine
Locations (1):
- Texas Children's Hospital Fetal Center and Newborn Center, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Keswani SG, Balaji S, Le LD, Leung A, Parvadia JK, Frischer J, Yamano S, Taichman N, Crombleholme TM. Role of salivary vascular endothelial growth factor (VEGF) in palatal mucosal wound healing. Wound Repair Regen. 2013 Jul-Aug;21(4):554-62. doi: 10.1111/wrr.12065. Epub 2013 Jun 11. PMID 23758212
- [Background] Section on Breastfeeding. Breastfeeding and the use of human milk. Pediatrics. 2012 Mar;129(3):e827-41. doi: 10.1542/peds.2011-3552. Epub 2012 Feb 27. PMID 22371471
- [Background] Rodriguez NA, Meier PP, Groer MW, Zeller JM. Oropharyngeal administration of colostrum to extremely low birth weight infants: theoretical perspectives. J Perinatol. 2009 Jan;29(1):1-7. doi: 10.1038/jp.2008.130. Epub 2008 Sep 4. PMID 18769379
- [Background] Gephart SM, Weller M. Colostrum as oral immune therapy to promote neonatal health. Adv Neonatal Care. 2014 Feb;14(1):44-51. doi: 10.1097/ANC.0000000000000052. PMID 24472888
- [Background] Rodriguez NA, Vento M, Claud EC, Wang CE, Caplan MS. Oropharyngeal administration of mother's colostrum, health outcomes of premature infants: study protocol for a randomized controlled trial. Trials. 2015 Oct 12;16:453. doi: 10.1186/s13063-015-0969-6. PMID 26458907
- [Background] Lee J, Kim HS, Jung YH, Choi KY, Shin SH, Kim EK, Choi JH. Oropharyngeal colostrum administration in extremely premature infants: an RCT. Pediatrics. 2015 Feb;135(2):e357-66. doi: 10.1542/peds.2014-2004. PMID 25624376
- [Background] Thibeau S, Boudreaux C. Exploring the use of mothers' own milk as oral care for mechanically ventilated very low-birth-weight preterm infants. Adv Neonatal Care. 2013 Jun;13(3):190-7. doi: 10.1097/ANC.0b013e318285f8e2. PMID 23722491
- [Background] Rodriguez NA, Caplan MS. Oropharyngeal administration of mother's milk to prevent necrotizing enterocolitis in extremely low-birth-weight infants: theoretical perspectives. J Perinat Neonatal Nurs. 2015 Jan-Mar;29(1):81-90. doi: 10.1097/JPN.0000000000000087. PMID 25633403
- [Background] McCallie KR, Lee HC, Mayer O, Cohen RS, Hintz SR, Rhine WD. Improved outcomes with a standardized feeding protocol for very low birth weight infants. J Perinatol. 2011 Apr;31 Suppl 1:S61-7. doi: 10.1038/jp.2010.185. PMID 21448207
- [Background] Seigel JK, Smith PB, Ashley PL, Cotten CM, Herbert CC, King BA, Maynor AR, Neill S, Wynn J, Bidegain M. Early administration of oropharyngeal colostrum to extremely low birth weight infants. Breastfeed Med. 2013 Dec;8(6):491-5. doi: 10.1089/bfm.2013.0025. Epub 2013 Jun 27. PMID 23805944
- [Background] Rodriguez NA, Meier PP, Groer MW, Zeller JM, Engstrom JL, Fogg L. A pilot study to determine the safety and feasibility of oropharyngeal administration of own mother's colostrum to extremely low-birth-weight infants. Adv Neonatal Care. 2010 Aug;10(4):206-12. doi: 10.1097/ANC.0b013e3181e94133. PMID 20697221
- [Background] Spinelli M, Frigerio A, Montali L, Fasolo M, Spada MS, Mangili G. 'I still have difficulties feeling like a mother': The transition to motherhood of preterm infants mothers. Psychol Health. 2016;31(2):184-204. doi: 10.1080/08870446.2015.1088015. Epub 2015 Oct 8. PMID 26359768
- [Background] Durfee SM, Benson CB, Adams SR, Ecker J, House M, Jennings R, Katz D, Pettigrew C, Wolfberg A. Postnatal outcome of fetuses with the prenatal diagnosis of gastroschisis. J Ultrasound Med. 2013 Mar;32(3):407-12. doi: 10.7863/jum.2013.32.3.407. PMID 23443180
- [Background] O'Connell RV, Dotters-Katz SK, Kuller JA, Strauss RA. Gastroschisis: A Review of Management and Outcomes. Obstet Gynecol Surv. 2016 Sep;71(9):537-44. doi: 10.1097/OGX.0000000000000344. PMID 27640608
- [Background] Gamba P, Midrio P. Abdominal wall defects: prenatal diagnosis, newborn management, and long-term outcomes. Semin Pediatr Surg. 2014 Oct;23(5):283-90. doi: 10.1053/j.sempedsurg.2014.09.009. Epub 2014 Sep 4. PMID 25459013
- [Background] Shah SK, Aroom KR, Walker PA, Xue H, Jimenez F, Gill BS, Cox CS Jr, Moore-Olufemi SD. Effects of nonocclusive mesenteric hypertension on intestinal function: implications for gastroschisis-related intestinal dysfunction. Pediatr Res. 2012 Jun;71(6):668-74. doi: 10.1038/pr.2012.20. Epub 2012 Feb 14. PMID 22476046
- [Background] Dalton BG, Gonzalez KW, Reddy SR, Hendrickson RJ, Iqbal CW. Improved outcomes for inborn babies with uncomplicated gastroschisis. J Pediatr Surg. 2017 Jul;52(7):1132-1134. doi: 10.1016/j.jpedsurg.2016.12.003. Epub 2016 Dec 18. PMID 28017414
- [Background] Hook-Dufresne DM, Yu X, Bandla V, Imseis E, Moore-Olufemi SD. The economic burden of gastroschisis: costs of a birth defect. J Surg Res. 2015 May 1;195(1):16-20. doi: 10.1016/j.jss.2015.01.036. Epub 2015 Jan 28. PMID 25703160
- [Background] Sydorak RM, Nijagal A, Sbragia L, Hirose S, Tsao K, Phibbs RH, Schmitt SK, Lee H, Farmer DL, Harrison MR, Albanese CT. Gastroschisis: small hole, big cost. J Pediatr Surg. 2002 Dec;37(12):1669-72. doi: 10.1053/jpsu.2002.36689. PMID 12483626
- [Background] Balgi S, Singhal S, Mueller G, Batton B. Feeding Intolerance and Poor Growth in Infants with Gastroschisis: Longitudinal Experience with Consecutive Patients over Thirteen Years. J Neonatal Surg. 2015 Oct 1;4(4):42. eCollection 2015 Oct-Dec. PMID 26500852
- [Background] Lao OB, Healey PJ, Perkins JD, Reyes JD, Goldin AB. Outcomes in children with intestinal failure following listing for intestinal transplant. J Pediatr Surg. 2010 Jan;45(1):100-7; discussion 107. doi: 10.1016/j.jpedsurg.2009.10.019. PMID 20105588
- [Background] Patel P, Bhatia J. Total parenteral nutrition for the very low birth weight infant. Semin Fetal Neonatal Med. 2017 Feb;22(1):2-7. doi: 10.1016/j.siny.2016.08.002. Epub 2016 Aug 27. PMID 27576106
- [Background] Stevens TP, Schulman J. Evidence-based approach to preventing central line-associated bloodstream infection in the NICU. Acta Paediatr. 2012 Apr;101(464):11-6. doi: 10.1111/j.1651-2227.2011.02547.x. PMID 22404886
- [Background] Mahieu LM, De Muynck AO, Ieven MM, De Dooy JJ, Goossens HJ, Van Reempts PJ. Risk factors for central vascular catheter-associated bloodstream infections among patients in a neonatal intensive care unit. J Hosp Infect. 2001 Jun;48(2):108-16. doi: 10.1053/jhin.2001.0984. PMID 11428877
- [Background] Squires RH, Duggan C, Teitelbaum DH, Wales PW, Balint J, Venick R, Rhee S, Sudan D, Mercer D, Martinez JA, Carter BA, Soden J, Horslen S, Rudolph JA, Kocoshis S, Superina R, Lawlor S, Haller T, Kurs-Lasky M, Belle SH; Pediatric Intestinal Failure Consortium. Natural history of pediatric intestinal failure: initial report from the Pediatric Intestinal Failure Consortium. J Pediatr. 2012 Oct;161(4):723-8.e2. doi: 10.1016/j.jpeds.2012.03.062. Epub 2012 May 11. PMID 22578586
- [Background] Miranda da Silva Alves F, Miranda ME, de Aguiar MJ, Bouzada Viana MC. Nutritional management and postoperative prognosis of newborns submitted to primary surgical repair of gastroschisis. J Pediatr (Rio J). 2016 May-Jun;92(3):268-75. doi: 10.1016/j.jped.2015.07.009. Epub 2016 Feb 2. PMID 26844392
- [Background] Aljahdali A, Mohajerani N, Skarsgard ED; Canadian Pediatric Surgery Network (CAPSNet). Effect of timing of enteral feeding on outcome in gastroschisis. J Pediatr Surg. 2013 May;48(5):971-6. doi: 10.1016/j.jpedsurg.2013.02.014. PMID 23701769
- [Background] Gulack BC, Laughon MM, Clark RH, Burgess T, Robinson S, Muhammad A, Zhang A, Davis A, Morton R, Chu VH, Arnold CJ, Hornik CP, Smith PB. Enteral Feeding with Human Milk Decreases Time to Discharge in Infants following Gastroschisis Repair. J Pediatr. 2016 Mar;170:85-9. doi: 10.1016/j.jpeds.2015.11.046. Epub 2015 Dec 15. PMID 26703875
- [Background] Torrazza RM, Neu J. The altered gut microbiome and necrotizing enterocolitis. Clin Perinatol. 2013 Mar;40(1):93-108. doi: 10.1016/j.clp.2012.12.009. PMID 23415266
- [Background] Min YW, Rhee PL. The Role of Microbiota on the Gut Immunology. Clin Ther. 2015 May 1;37(5):968-75. doi: 10.1016/j.clinthera.2015.03.009. Epub 2015 Apr 4. PMID 25846321
- [Background] Neu J, Pammi M. Pathogenesis of NEC: Impact of an altered intestinal microbiome. Semin Perinatol. 2017 Feb;41(1):29-35. doi: 10.1053/j.semperi.2016.09.015. Epub 2016 Dec 13. PMID 27986328
- [Background] Westerbeek EA, van den Berg A, Lafeber HN, Knol J, Fetter WP, van Elburg RM. The intestinal bacterial colonisation in preterm infants: a review of the literature. Clin Nutr. 2006 Jun;25(3):361-8. doi: 10.1016/j.clnu.2006.03.002. Epub 2006 May 4. PMID 16677741
- [Background] Liu S. The Development of Our Organ of Other Kinds-The Gut Microbiota. Front Microbiol. 2016 Dec 23;7:2107. doi: 10.3389/fmicb.2016.02107. eCollection 2016. No abstract available. PMID 28066404
- [Background] Meropol SB, Edwards A. Development of the infant intestinal microbiome: A bird's eye view of a complex process. Birth Defects Res C Embryo Today. 2015 Dec;105(4):228-39. doi: 10.1002/bdrc.21114. Epub 2015 Dec 11. PMID 26663826
- [Background] Magne F, Suau A, Pochart P, Desjeux JF. Fecal microbial community in preterm infants. J Pediatr Gastroenterol Nutr. 2005 Oct;41(4):386-92. doi: 10.1097/01.mpg.0000179855.38543.85. No abstract available. PMID 16205503
- [Background] Sohn K, Kalanetra KM, Mills DA, Underwood MA. Buccal administration of human colostrum: impact on the oral microbiota of premature infants. J Perinatol. 2016 Feb;36(2):106-11. doi: 10.1038/jp.2015.157. Epub 2015 Dec 10. PMID 26658119